CLINICAL TRIAL: NCT04195620
Title: The Role of Vulnerability and Responsiveness in Cardiovascular Disease Biomarkers Associated With Loneliness
Brief Title: Loneliness and Social Connection in Cardiovascular Disease
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: University affiliation changed and I was unable to transfer the grant that was funding the project
Sponsor: Morehead State University (Other)
Responsible Party: Principal Investigator, Daniel Maitland, Assistant Professor of Psychology, Morehead State University
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Other
Other Study IDs: HRVLoneliness
Record Dates: First submitted 2019-12-10; First posted 2019-12-12 (Actual); Last update posted 2022-04-29 (Actual); Status verified 2022-04

CONDITIONS: Cardiovascular Diseases
Keywords: Loneliness; Sympathetic Nervous System; Parasympathetic Nervous System; Vulnerability; Self-disclosure
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Intervention Model Description: 2x2 factorial design assessing different levels of loneliness and those individuals being randomized to one of two conditions involving either high levels of self-disclosure or low levels of self-dislcosure
Who Masked: Investigator
Masking Description: The investigator will be naïve to participant treatment condition. All other individuals will know or it will be obvious to them.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Low loneliness, low self-disclosure (Experimental): Individuals in this arm report lower levels of loneliness than the mean level reported by similar individuals. They will start the study in the low self-disclosure group which involves questions that are unlikely to involve meaningful personal disclosure. All members of this group will also complete the high self-disclosure condition later in the study.
  Interventions: Other: High self-disclosure; Other: Low self-disclosure
- Low loneliness, high self-disclosure (Experimental): Individuals in this arm report lower levels of loneliness than the mean level reported by similar individuals. They will start the study in the high self-disclosure group which involves questions that are likely to involve meaningful personal disclosure. All members of this group will also complete the low self-disclosure condition later in the study.
  Interventions: Other: High self-disclosure; Other: Low self-disclosure
- high loneliness, low self-disclosure (Experimental): Individuals in this arm report higher levels of loneliness than the mean level reported by similar individuals. They will start the study in the low self-disclosure group which involves questions that are unlikely to involve meaningful personal disclosure. All members of this group will also complete the high self-disclosure condition later in the study.
  Interventions: Other: High self-disclosure; Other: Low self-disclosure
- high loneliness, high self-disclosure (Experimental): Individuals in this arm report higher levels of loneliness than the mean level reported by similar individuals. They will start the study in the high self-disclosure group which involves questions that are likely to involve meaningful personal disclosure. All members of this group will also complete the low self-disclosure condition later in the study.
  Interventions: Other: High self-disclosure; Other: Low self-disclosure

INTERVENTIONS:
Other: High self-disclosure — The high self-disclosure condition involves individuals asking and answering a series of questions that are more personal in nature and involve sharing or receiving information that is likely to be emotionally laden and information that is not readily shared in typical conversations. An example of a question from this condition includes "If you were to die today without the chance to speak with anyone, what would you most regret not having said to someone? Why haven't you said it yet?"
Other: Low self-disclosure — The low self-disclosure condition involves individuals asking and answering a series of questions that are not personal in nature and involve sharing or receiving information that is shared in very casual conversations. An example of a question from this condition includes "What did you do to celebrate Halloween last year?"

SUMMARY:
The study evaluates the impact of vulnerable self-disclosure and perceived responsiveness in individuals across levels of loneliness. Participants will be randomized to a high disclosure or a low disclosure condition.

DETAILED DESCRIPTION:
Recent studies have found that loneliness has the same impact on morbidity and mortality as smoking cigarettes and twice that of obesity. One proposed pathway by which loneliness impacts morbidity and mortality is through cardiovascular disease. Loneliness is regularly associated with increased sympathetic nervous system and decreased parasympathetic nervous system engagement, both reliable biomarkers of increased risk of cardiovascular disease. One possible explanation for the this phenomena is that individuals who experience loneliness experience meaningful disruptions to the interpersonal process where they fail to disclose when appropriate or react to other individuals disclosure. This may result in engagement of nervous system regulation of social behaviors resulting in both in the moment and long term engagement of the sympathetic nervous system. The proposed 2-year research plan will examine the behaviors and nervous system reactions of individuals across loneliness levels in an experimental condition that manipulates the probability of engaging in relationship building behaviors.

This study will recruit 60 individuals aged 18-25 who are fluent in English and report no history of cardiovascular or respiratory disease to participate in a study investigating social interactions. While a specific level of loneliness is not an inclusion variable, to ensure representation across loneliness levels, the investigators will screen for levels of loneliness and invite individuals to participate equally distributed between 4 levels of loneliness: 1 or more standard deviations below the mean, between 0-1 standard deviations below the mean, between 0-1 standard deviations above the mean, and 1 standard deviation or more above the mean.

The study will then utilize a 2x2 factorial design splitting participants into reporting above or below the mean level of loneliness and randomizing those individuals to a behavioral task condition that involves answering either a high disclosure or low disclosure set of questions. Before engaging in the behavioral task, participants will fill out a series of questionnaires assessing their current social functioning. Participants will then have baseline levels of sympathetic nervous system and parasympathetic nervous system engagement measured. In an ongoing way, throughout the behavioral task, participants will have their of sympathetic nervous system and parasympathetic nervous system engagement measured. Every 15 minutes, the behavioral task will stop and participants will complete a series of questionnaires assessing their evaluation of their behavior with the research assistant in the task, as well as feelings of connection they are experiencing with the research assistant. At the conclusion of the behavioral task, participants will be invited back to participate in the condition they had not previously completed with a new research assistant. All behavioral tasks will be coded by trained research assistants assessing third party evaluation of relationship building behaviors.

ELIGIBILITY:
Inclusion Criteria:

* Being between the ages (inclusive) of 18-25
* English as a primary language
* Provides consent

Exclusion Criteria:

* Known heart condition
* Known respiratory condition
* Inability to transport themselves to and from Morehead State University's campus

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 34 (Actual)
Dates: Start 2020-09-01 (Actual); Primary Completion 2022-01-01 (Actual); Study Completion 2022-01-01 (Actual)

PRIMARY OUTCOMES:
Respiratory Sinus Arrhythmia | 50 minutes
  Respiratory sinus arrhythmia (RSA) is heart rate variability in synchrony with respiration. RSA is considered a reliable way to measure parasympathetic innervation of the heart mediated by the vagus nerve.
Electrodermal Activity | 50 minutes
  Electrodermal activity (EDA) is the property of the body that results in variation in the electrical characteristics of the skin. It is thought that skin resistance varies as a function of the state of sweat glands in the skin and that sweating is controlled by the sympathetic nervous system. Consequently, EDA is viewed as a non-invasive measure of sympathetic nervous system activity.

SECONDARY OUTCOMES:
Self-reported Feelings of Connection | 50 minutes
  The Social Connectedness Scale: Research Assistant. The minimum score on the measure is 6, the maximum is 36. Higher scores on the measure indicate more feelings of connection. The measure is a composite of 6 questions assessing feelings of connection reported by the participant. All 6 questions are measured on a scale of 1-6.

CONTACTS AND LOCATIONS:
Locations (1):
- Morehead State University, Morehead, Kentucky, United States

IPD SHARING:
Plan to Share IPD: Yes
Given that the data collected contains no identifiers, all IPD will be made available.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Pending completion of data collection and cleaning.
URL: https://cos.io/